CLINICAL TRIAL: NCT06494813
Title: Biochemical Role of Matrix Metalloproteinase -9 in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Basma Aboelfotoh Mahmoud, demonstrator of medical biochemistry, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med-24-06-08MS
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controls (Active Comparator): apparently healthy individual with no chronic illness
  Interventions: Diagnostic Test: conventional pcr
- cases (Active Comparator): patients with rheumatoid arthritis who fulfilled the EULAR/ACR Criteria 2010 for the Classification of RA
  Interventions: Diagnostic Test: conventional pcr

INTERVENTIONS:
Diagnostic Test: conventional pcr — conventional pcr to study matrix metalloproteinase -9 gene polymorphismin rheumatoid arthritis

SUMMARY:
Rheumatoid arthritis (RA) is a systemic autoimmune pathology associated with a chronic inflammatory process, which can damage both joints and extra-articular organs, including the heart, kidney, lung, digestive system, eye, skin and nervous system.(Cojocaru et al. 2010, Conforti et al. 2021).

Rheumatoid arthritis affects most commonly the hand, wrist, and foot, but it can also affect large joints .IT is characterized by painful, swollen joints that can severely impair physical function and quality of life and associated with increased mortality (Sparks et al. 2016). About 70% of patients with RA are women, and peak incidence is between ages 50 and 60 years (Sparks et al. 2019).

Matrix Metalloproteinases are a family of calcium-dependent endopeptidases with a zinc-binding active side. More than 20 different MMPs are classified according to the particular substrates they degrade: collagenases, stromelysins, gelatinases, matrilysins, membrane-type MMPs, and others. Moreover, MMPs release growth factors from carrier proteins, inactivate proteinase inhibitors, and influence inflammatory cytokines and chemokines that can also be responsible for joint destruction(Nagase et al. 2006) .

In the human body, MMPs are synthesized in leukocytes, macrophages, endothelial cells, and connective tissue cells such as chondrocytes and synoviocytes, both found in the knee joint. Matrix metalloproteinases are secreted as pre-proenzymes into the extracellular fluid, where they can be activated by a variety of substances: epidermal growth factor (EGF), vascular endothelial growth factor (VEGF), tumor necrosis factor-α (TNF-α), interleukin-1 (IL-1), and other MMPs. Conversely, steroid hormones, transforming growth factor-β (TGF-β), plasma proteins such as a2-macroglobulin and a1-antitrypsin, and tissue inhibitors of metalloproteinases (TIMPs) can inhibit MMP activity(Visse and Nagase 2003).

The pathogenesis of RA is based on the fact that the patient's body reacts to autoantigens, e.g. citrullinated peptides, or a foreign peptide, e.g. a viral or bacterial peptide that is cross-reactive with an autoantigen (Kwon and Ju 2021).

Activated T cells, B cells, and monocytes infiltrate the synovial membrane in joints, as that is where the autoantigens accumulate. Cytokines and chemokines secreted by leukocytes, such as tumor necrosis factor, IL-6, and granulocyte colony-stimulating factors activate endothelial cells, stimulate neovascularization and leukocyte migration, and cause expansion of synovial fibroblast-like and macrophage-like cells (Alivernini et al. 2022). Expansion of these cells leads to a hyperplastic synovial lining layer referred to as a "pannus". The pannus invades the periarticular bone at the cartilage-bone junction and leads to the progressive destruction of cartilage and subchondral bone tissue(Aletaha and Smolen 2018).

Matrix metalloproteinases are crucial for the pathogenesis of RA. Synovial fibroblast-like cells, having a tumor-like appearance, secrete various proteases, including MMPs that degrade ECM components, mainly proteoglycans, and collagens, of articular cartilage in the affected joints. Expression of the following MMPs is upregulated in synovial tissue: MMP-1, -3, -9, and -13 (Vincenti and Brinckerhoff 2002, Heard et al. 2012, Araki and Mimura 2017).

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis who fulfilled the EULAR/ACR Criteria 2010 for the Classification of RA .. All patients recruited for the study had active RA confirmed by assessment of activity by DAS28 .

Exclusion Criteria:

* No patient had a history of tuberculosis or symptoms of infectious diseases in the previous 3 months.

2-30 healthy subjects; age and sex mateched to the patients as healthy controls.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
matrix metalloproteinase -9 gene poly morphism | 12 months
  matrix metalloproteinase -9 gene poly morphism quantification by conventional pcr

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aletaha D, Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018 Oct 2;320(13):1360-1372. doi: 10.1001/jama.2018.13103. PMID 30285183
- [Background] Araki Y, Mimura T. Matrix Metalloproteinase Gene Activation Resulting from Disordred Epigenetic Mechanisms in Rheumatoid Arthritis. Int J Mol Sci. 2017 Apr 25;18(5):905. doi: 10.3390/ijms18050905. PMID 28441353
- [Background] Alivernini S, Firestein GS, McInnes IB. The pathogenesis of rheumatoid arthritis. Immunity. 2022 Dec 13;55(12):2255-2270. doi: 10.1016/j.immuni.2022.11.009. PMID 36516818
- [Background] Cojocaru M, Cojocaru IM, Silosi I, Vrabie CD, Tanasescu R. Extra-articular Manifestations in Rheumatoid Arthritis. Maedica (Bucur). 2010 Dec;5(4):286-91. PMID 21977172